CLINICAL TRIAL: NCT04343911
Title: Position-related Postoperative Peripheral Neuropathy After Laparoscopic Colorectal Surgery - a Comparative Single-center Prospective Cohort Study
Brief Title: Postoperative Peripheral Neuropathy After Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Signe Amalie Wolthers Laursen, Principal Investigator and Specialist Registrar in Anesthesiology, Copenhagen University Hospital, Hvidovre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 44954
Record Dates: First submitted 2020-02-13; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Peripheral Neuropathy; Postoperative Complications
Keywords: positioning; neuropathy; trendelenburg
MeSH Terms: conditions — Peripheral Nervous System Diseases; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional positioning (No Intervention): positioning with shoulder braces
- positioning on Pink Pad ® (Active Comparator)
  Interventions: Device: Pink Pad ® (Xodus Medical Inc., New Kensington, PA)

INTERVENTIONS:
Device: Pink Pad ® (Xodus Medical Inc., New Kensington, PA) — a non-sliding foam mattress
  Arms: positioning on Pink Pad ®

SUMMARY:
This prospective cohort study of patients undergoing colorectal surgery positioned conventionally with shoulder braces was performed. After initial results the implementation of the Pink Pad ® took place in order to compare the two groups. This study favours Pink Pad over conventional positioning concerning postoperative neuropathy.

DETAILED DESCRIPTION:
Laparoscopic colorectal surgery requires perioperative positioning in the dorsal lithotomy position and intermittent Trendelenburg position, which is associated with postoperative peripheral neuropathy, which is a substantial cause of anesthesia-related claims. This study aims to primarily assess the incidence of postoperative peripheral neuropathy of patients positioned conventionally by shoulder braces and secondly to compare this group with patients positioned on the foam mattress Pink Pad ® 24-hours after surgery and secondarily at a 30-day postoperative follow-up.

This consecutive single-center prospective cohort study of 155 patients undergoing colorectal surgery was performed between November 2014 and June 2015. After initial results the implementation of the Pink Pad ® took place and a total of 52 patients were included between May 2016 and February 2017 in order to compare the two groups.

Position related postoperative peripheral neuropathy is an important complication after laparoscopic colorectal surgery. This study concludes that careful attention should be payed to positioning and favors Pink Pad ® over conventional positioning with shoulder braces.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Elective laparoscopic colorectal surgery
* Sufficient written and verbal Danish skills
* Awake, responsive and oriented in the post-surgical inclusion period

Exclusion Criteria:

* Pre-existing peripheral neuro- or musculopathy,
* Conversion to open operation
* Lack of consent were defined as exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
position related postoperative peripheral neuropathy | 24-hours after surgery
  This study's primary outcome is to evaluated the incidence of postoperative peripheral neuropathy in patients positioned conventionally compared to patients positioned on the Pink Pad foam mattress 24-hours after surgery.

SECONDARY OUTCOMES:
Position related postoperative peripheral neuropathy | 30 day follow-up after surgery
  The secondary outcome of this study is to evaluate the incidence of postoperative peripheral neuropathy in patients positioned conventionally compared to patients positioned on the Pink Pad foam mattress 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Signe AW Laursen, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No